CLINICAL TRIAL: NCT04990570
Title: Telemedicine (Virtual Clinic) Effectively Delivers the Required Health-care Service for Pediatric Day-case Surgical Patients in the Current Era of Covid -19 Pandemic: A Non-randomized Controlled Study
Brief Title: Telemedicine (Virtual Clinic) for Pediatric Surgery During Covid-19 Pandemic
Acronym: TelemedCov
Status: Completed | Type: Observational
Sponsor: dr. Muhammad Abdelhafez Mahmoud, MD (Other)
Responsible Party: Sponsor-Investigator, dr. Muhammad Abdelhafez Mahmoud, MD, Lecturer of pediatric surgery, Al-Azhar Faculty of Medicine, Al-Azhar University
Organization: Al-Azhar University (Other)
Other Study IDs: Al-AzharTelemedicineinCovid-19
Record Dates: First submitted 2021-08-02; First posted 2021-08-04 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Telemedicine; Virtual Clinic; Covid19; Pandemic
Keywords: Telemedicine;; Covid-19 Pandemic;; Pediatric Surgery;; Children;; Video Conversation;; Patient's Privacy;; Data Security; Health-care Service; Day-case Surgery
MeSH Terms: conditions — COVID-19 | interventions — Telemedicine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pediatric day-case surgical patients, encountered via Virtual clinic from June 2020 till July 2021: Pediatric patients, with age ranging from 1 month-14 years, with day-case surgical problems, encountered during the era of Covid-19 pandemic.
  Telemedicine, in the form of Virtual clinic, was utilized to address this distressing problem, to aid in conveying their concerns and bridge the gap in surgeon-patient relationship & encounter.
  Interventions: Other: Telemedicine in the form Virtual clinic via video consultation
- Control group comprising of patients scheduled to the OPD clinic from June 2019 till June 2020: Cases of office OPD appointments in the period from June 2019 till June 2020 will be included as a control group

INTERVENTIONS:
Other: Telemedicine in the form Virtual clinic via video consultation — Pediatric patients, with age ranging from 1 month-14 years, with surgical problems, encountered during the era of Covid-19 pandemic.
  Some of them seen at the OPD clinic, while the majority failed to attend because of Covid-19 associated lock-down and Curfew, thus, rendering their approach to the service.
  Telemedicine, in the form of Virtual clinic, was utilized to address the distressing problem of difficult approach of patients to the pedia surgery OPD because of Covid-19 pandemic restrictive regulatory precautions, to aid in conveying their concerns and bridge the gap in surgeon-patient relationship & encounter.
  Groups: Pediatric day-case surgical patients, encountered via Virtual clinic from June 2020 till July 2021

SUMMARY:
Telemedicine (Virtual Clinic) Effectively Delivers the Required Health-care Service to Pediatric Day-case Surgical Patients in the Current Era of Covid-19 Pandemic: A Non-randomized Controlled Study

DETAILED DESCRIPTION:
Children often get sick, either from congenital or acquired lesions. The Covid-19 associated regulatory precautions had made the process of seeking medical advice getting more difficult and much challenging. In this article, we aim to present our experience in utilization of telemedicine, specifically the virtual clinic via video consultation, in sorting and guiding the pediatric surgical patients, evaluate the effectiveness, and document its results in giving a convenient solution for this heavily distressing problem.

Materials and Methods:

This prospective study addressed the utilization of telemedicine, specifically the virtual clinic via video consultation in the field of pediatric surgery in the current era of Covid-19 pandemic. Data recorded for analysis included demographic data, condition distribution (system/body region affected), conversation duration, ultimate fate of the consultations. Service was evaluated by on-line patient questionnaire ranging from 1 to 5.

Study was carried out at 3 pediatric surgery tertiary centers (Prince Mohammed bin Abdulaziz Hospital in Riyadh, Alyamamah Obstetric & Children's hospital in Riyadh, and Al-Azhar University hospitals in Cairo) on pediatric surgical patients, in the period from June 2020 to July 2021, in comparison to the statistics of the period from June 2019 till June 2020. All patients' guardians enrolled in the study had electronically signed a written informed consent before commencement of a video consultation. The study was approved by the Institutional Review Board and ethics committee (Registration number: H7D4-2020-0051E). The main objective was to assess the efficacy utilization of telemedicine (mainly virtual clinic via video consultation) in sorting and correct guiding of children with surgical issues. Primary outcome measurements included attendance rate, cancellation rate, re-admission rate, and parent/patients' satisfaction. Secondary outcome measurements included time interval from appointment request till the actual encounter, encounter duration, and fate of the video conversations.

All patients are requested to register in the MOH registry (including ID and phone numbers, address, & e-mail), and are given instructions on how to use the certified applications to organize their access to the service via approved applications at any time. Also, on-call pediatric surgery specialists were ready all the time.

Telemedicine (virtual clinic via video consultation), between a well-trained expert pediatric surgeon and a motivated child's caregiver, effectively bridges the gap caused by the regulatory precautions mandated by the current Covid-19 pandemic.

Statistical analysis:

It will be performed with IBM SPSS Statistics for Windows, Version 23.0. Armonk, NY: IBM Corp. Data will be presented as mean, standard deviation, number & percentage, using Chi-squared test (X2) for qualitative data. The significance level will be set at P > 0.05.

- Discussion will focus on demonstrating and achieving the main objective that was to assess the efficacy utilization of telemedicine (mainly virtual clinic via video consultation) in sorting and correct guiding of children with surgical issues. Points of discussion will include attendance rate, cancellation rate, re-admission rate, and parent/patients' satisfaction, fate of the video conversations.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients, with surgical conditions or consultations
* Mindful parents, motivated to use this remote interaction technology
* Available equipment (smart phone, computer or laptop, or tablet and strong stable internet connection with Ethernet coverage)

Exclusion Criteria:

* Patients older than 14 yrs of age
* Parents/patients refuse this method of interaction
* Equipment shortage
* Poor internet connection

Ages: 1 Month to 14 Years | Sex: All
Age Groups: Child
Study Population: Pediatric surgical patients, with age ranging from 1 month till 14 yrs old, in need to surgical consultation and further management of their issues in the era of Covid-19 pandemic, with the majority being rendered from approach to the OPD because of Covid-19 associated regulatory precautions notably lockdown period and Curfew
Sampling Method: Non-Probability Sample
Enrollment: 1396 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-06-07 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Age of patients | 1 year
  Age in years
Condition distribution | 1 year
  Condition distribution in percentage
Conversation duration | 1 year
  Conversation duration in minutes
Attendance rate | 1 year
  Attendance rate in percentage
Cancellation rate | 1 year
  Cancellation rate in percentage
Rate of re-admissions | 1 year
  Rate of re-admissions in percentage

SECONDARY OUTCOMES:
Ultimate fate of the interview | 1 year
  Ultimate fate of the interview in ratio
Patient satisfaction questionnaire | 1 year
  Patient satisfaction degree in numbers

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Elsayed AH Mahmoud, MD, Principal Investigator — Al-Azhar University, Faculty of Medicine
Locations (1):
- Muhammad Elsayed Abdelhafez Mahmoud, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Data are available for other researchers including methodology, figures, tables, results, and philosophy of discussion and the value this study add to the literature
Supporting Information: Study Protocol, SAP, ICF
Time Frame: August 2021 till indefinitely
Access Criteria: Send a request to the study principal-investigator
URL: http://orcid.org/0000-0002-6328-6419